CLINICAL TRIAL: NCT01051921
Title: An Open-Label Trial of Pegylated Interferon Plus Ribavirin in Combination With CTS-1027 in HCV Null-Responders
Brief Title: Study of CTS-1027 in Combination With Pegylated Interferon and Ribavirin in Hepatitis C Virus (HCV) Null-Responders
Acronym: CTS-1027-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTS-1027-04
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis C
Keywords: HCV; Null Responder
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CTS-1027, Peg IFN, Ribavirin (Experimental): Study drug (CTS-1027) plus Standard of Care treatment (pegylated interferon and ribavirin).
  CTS-1027, 15 mg taken twice daily. Pegylated interferon, 180 μg injected once a week. Ribavirin, 1000 mg or 1200 mg daily (depending on patient weight), taken in two divided doses.
  Interventions: Drug: CTS-1027; Drug: Pegylated interferon; Drug: Ribavirin

INTERVENTIONS:
Drug: CTS-1027 — CTS-1027 supplied in 5 and 10 mg tablets, 15 mg taken twice daily, for up to 48 weeks
Drug: Pegylated interferon — Pegylated interferon, 180 micrograms in 0.5 ml of solution injected subcutaneously (SQ) once per week, for up to 48 weeks. Packaged in single use syringes.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin, 200 mg capsules taken in two divided daily doses totaling 1000 mg (5 capsules) for patients weighing 75 kg or less, or 1200 mg (6 capsules) for patients weighing more than 75 kg for up to 48 weeks.
  Other Names: Copegus

SUMMARY:
The purpose of this study is to determine if the combination treatment of CTS-1027, pegylated interferon and ribavirin can improve the response rates in HCV patients who did not previously respond to pegylated interferon and ribavirin therapy.

DETAILED DESCRIPTION:
A subset of non-responders to standard of care treatments (pegylated interferon and ribavrin) is termed null responders. Null responders are the most treatment refractory population. Treatment for null responders is currently limited: retreatment with SOC results in approximately 5% sustained virologic response (SVR).

CTS-1027 may facilitate the activity of interferon by preventing MMP-induced cleavage and deactivation in both phases of clinical response to therapy. In addition, CTS-1027, like ribavirin, alone does not significantly affect viral replication, but both CTS-1027 and ribavirin are likely to impact response to therapy during the second and slower phase of the clinical response.

The potential of MMP inhibition to facilitate the action of interferon, together with ribavirin-driven up-regulation of interferon stimulated genes, has the potential to yield a potent host immune response in this highly resistant null-responder patient population. Again, since MMP inhibition is thought to target the second slower phase kinetics, the initial treatment duration in this trial will be 24 weeks.

This trial will evaluate the safety and efficacy of CTS-1027 combined with SOC in patients who did not previously respond to SOC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the trial
* HCV genotype 1 infected null responders to prior therapy comprised of pegylated interferon and ribavirin (standard of care, SOC) defined as:

  * Failure to achieve an early virologic response (< 2 log decline in HCV-RNA by Week 12), or
  * If Week 12 HCV-RNA was not obtained but Week 24 was obtained, Week 24 response was < 2 log decline
* Alpha-fetoprotein (AFP) <= 50 ng/mL
* Hemoglobin ≥ 12 g/dL, platelet count ≥ 125 x 10^9/L, and white blood cell count ≥ 1.5 x 10^9/L
* In the opinion of the Principal Investigator, the patient met the 80%/80%/80% rule during the previous pegylated interferon and ribavirin therapy (i.e., received at least 80% of the pegylated interferon and ribavirin doses, at least 80% of the dose size, for at least 80% of the treatment duration)
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from screening to at least six months after the completion of the trial.

Exclusion Criteria:

* < 2 log decline in HCV-RNA at Week 12 but > 2 log decline at any time from Week 12 to Week 24 during prior therapy with pegylated interferon and ribavirin (prior standard of care therapy)
* Decompensated or severe liver disease defined by one or more of the following criteria:

  * Prothrombin time 3 seconds > control
  * Direct bilirubin ≥ 1.5 x ULN
  * Serum albumin below normal limits
  * AST or ALT > 7 x ULN at screening
* Evidence of portal hypertension including:

  * Varices on esophagogastroduodenoscopy (EGD) with or without a history of gastrointestinal bleeding; or
  * Ascites
* Cirrhosis defined by one or both of the following criteria:

  * Liver biopsy showing cirrhosis
  * Other clinical signs and symptoms suggestive of cirrhosis
* Hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound (or other imaging techniques)
* Clinically significant ocular findings such as retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or other abnormality
* Known history or presence of human immunodeficiency virus (HIV) infection
* Co-infection with hepatitis B virus (HBV)
* If female: pregnant, lactating, or positive serum or urine pregnancy test
* Male partners of women who are currently pregnant
* Renal impairment (creatinine > 1.5 x ULN), creatinine clearance < 50 mL/min, or hepatorenal syndrome with ascites
* Hospitalization for liver disease within 60 days of screening
* History of alcohol abuse (> 50 g per day) within the past year
* History of severe psychiatric disease, especially depression, characterized by:

  * Suicide attempt
  * Hospitalization for psychiatric disease
  * Period of disability as a result of psychiatric disease
* Prior exposure to CTS-1027
* Prior triple treatment comprised of pegylated interferon, ribavirin, and protease and/or polymerase inhibitors
* History or presence of clinically concerning cardiac arrhythmias or prolongation of pre-dose QTc interval of > 450 milliseconds
* Other concomitant disease or condition likely to significantly decrease life expectancy (e.g., moderate to severe congestive heart failure) or any malignancy other than curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for ten or more years
* Any patient who has received any investigational drug or device within 30 days of dosing, or who is scheduled to receive another investigational drug or device during the course of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Castelloe, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (15):
- United States (14):
  - Scripps Clinic, La Jolla, California
  - VA Medical Center, San Diego, San Diego, California
  - University of Colorado Health Science Center, Denver, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - MN Clinical Research Center, Plymouth, Minnesota
  - St. Louis University, St Louis, Missouri
  - Consultants of Clinical Research, Ohio GI and Liver Institute, Cincinnati, Ohio
  - Advanced Liver Therapies - Baylor College of Medicine, Houston, Texas
  - VA Medical Center, Houston, Houston, Texas
  - University of Utah Health Science Center, Salt Lake City, Utah
  - Liver Institute of Virginia, Newport News, Virginia
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- CTS-1027, Pegylated Interferon, Ribavirin: CTS-1027 plus Pegylated Interferon plus ribavirin
Period: Overall Study
Arm/Group | CTS-1027, Pegylated Interferon, Ribavirin
Started | 67
Completed | 37
Not Completed | 30
Not completed — Physician Decision | 9
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 4
Not completed — virological failure | 1
Not completed — patient moved | 1

BASELINE CHARACTERISTICS:
Arm/Group | CTS-1027, Pegylated Interferon, Ribavirin
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Early Virologic Response (EVR)
Description: Early Virologic Response (EVR) is defined as the percent of patients who experienced a drop in HCV-RNA (Hepatitis C Ribonucleic acid, also known as "viral load") levels of more that 2 log from before treatment (baseline) through 12 Weeks of treatment.
Time Frame: Baseline and Study week 12
Population: Although this study was completed, the entire CTS-1027 program was discontinued prior to database lock. Therefore, efficacy analysis was not completed for this study.
Measure: Number; unit: Percent of Patients
Groups:
- CTS-1027, Pegylated Interferon, Ribavirin: CTS-1027, 5mg and 10 mg tablets (one each) taken twice daily for a total daily dose of 30 mg.
  Pegylated Interferon, individual syringes delivering 180 µg of drug in 0.5 ml of solution administered once weekly.
  Ribavirin, 200 mg capsules, taken in two divided daily doses totaling 1000 mg (5 capsules) daily for patients weighing 75kg or less, and 1200 mg (6 capsules) daily for patients weighing more than 75 kg
Arm/Group | CTS-1027, Pegylated Interferon, Ribavirin
Number analyzed (Participants) | 0

2. Secondary Outcome: > 2 Log Decline in Hepatitis C Virus Ribonucleic Acid (HCV-RNA) at 24 Weeks
Description: Percent of patients experiencing a drop in HCV-RNA Hepatitis C virus ribonucleic acid, also known as "viral load") levels in the blood equal to, or greater than, 2 log from before treatment (baseline) through 24 weeks of treatment.
Time Frame: Baseline and Study week 24
Population: as for outcome 1
Measure: Number; unit: Percent of patients
Arm/Group | CTS-1027, Pegylated Interferon, Ribavirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing through 12 week follow-up visit (up to 60 weeks).
Description: Adverse events listed are those reported by at least 5% of the patients, and deemed potentially related (possibly, probably, or definitely) by the Investigator. All serious adverse events are reported regardless of causality.
Arm/Group | CTS-1027, Pegylated Interferon, Ribavirin
Serious Adverse Events (participants affected / at risk) | 7/67
Other Adverse Events (participants affected / at risk) | 63/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027, Pegylated Interferon, Ribavirin (N=67)
Appendicitis (Infections and infestations) | 1 (1)
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTS-1027, Pegylated Interferon, Ribavirin (N=67)
Anemia (Blood and lymphatic system disorders) | 18 (31)
Neutropenia (Blood and lymphatic system disorders) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 8 (11)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 9 (9)
Fatigue (General disorders) | 38 (62)
Influenza like illness (General disorders) | 8 (10)
Injection site reaction (General disorders) | 4 (4)
Irritability (General disorders) | 11 (17)
Pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 8 (11)
Sinusitis (Infections and infestations) | 4 (4)
Wieght decreased (Investigations) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (58)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (30)
Disturbance in attention (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 8 (9)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 24 (38)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 17 (25)
Insomnia (Psychiatric disorders) | 15 (24)
Mood swings (Psychiatric disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (18)
Rash (Skin and subcutaneous tissue disorders) | 10 (16)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (8)

LIMITATIONS AND CAVEATS:
Although this study was completed, the entire CTS-1027 program was discontinued prior to database lock. Hence, only a safety analysis was carried out for this study. Analysis of the primary and secondary efficacy measures was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less